CLINICAL TRIAL: NCT00147667
Title: Randomised Double Blind Placebo Controlled Trial of Effects of Long Term Low Dose Oral Erythromycin Therapy in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Long Term Macrolide Antibiotic Therapy in Patients With COPD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Free and University College Medical School (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P03/03
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2005-09-07 (Estimated); Status verified 2004-03

CONDITIONS: COPD
Keywords: COPD; EXACERBATIONS; AIRWAY INFLAMMATION
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Erythromycin

INTERVENTIONS:
Drug: Erythromycin

SUMMARY:
The purpose of this study is to determine whether long term treatment with oral erythromycin is effective in the treatment of subjects with Chronic Obstructive Pulmonary Disease (COPD) by reducing the number of exacerbations and the degree of airway inflammation.

DETAILED DESCRIPTION:
COPD is characterised by persisting airway inflammation which leads to a progressive and irreversible deterioration in lung function with the eventual development of respiratory symptoms which may become disabling. Periodic episodes of worsening symptoms or exacerbations are a major cause of additional morbidity, mortality and health care utilization. Currently available therapies have limited efficacy in reducing airway inflammation or preventing exacerbations.

Macrolides such as erythromycin have been shown to have potent anti-inflammatory effects in in vitro experiments and in other lung conditions such as cystic fibrosis and bronchiectasis as well as in open label studies in COPD. We hypothesised that long term therapy with oral erythromycin would reduce airway inflammation and reduce the frequency of exacerbations in patients with COPD. If these properties are demonstrated this therapy can have potentially important benefits if effective in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of COPD
* Clinically stable for 6 weeks
* Able to Swallow Tablets

Exclusion Criteria:

* Clinically significant respiratory disease other than COPD
* Women of child bearing age
* Patients receiving existing Medication which may interact adversely with trial drug
* History of clinically significant liver disease

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-04; Study Completion 2006-03

PRIMARY OUTCOMES:
Exacerbation Frequency
Airway Inflammation

SECONDARY OUTCOMES:
Lung Function
Health Status
Exacerbation Recovery Time
Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga A Wedzicha, MD, Principal Investigator — Royal Free and University College Medical School
Locations (1):
- Royal Free Hospital, London, England, United Kingdom

REFERENCES:
- [Derived] Seemungal TA, Wilkinson TM, Hurst JR, Perera WR, Sapsford RJ, Wedzicha JA. Long-term erythromycin therapy is associated with decreased chronic obstructive pulmonary disease exacerbations. Am J Respir Crit Care Med. 2008 Dec 1;178(11):1139-47. doi: 10.1164/rccm.200801-145OC. Epub 2008 Aug 21. PMID 18723437